CLINICAL TRIAL: NCT05281042
Title: Home OCT Repeatability and Reproducibility of Automatic Fluid Quantification Study
Status: Completed | Type: Observational
Sponsor: Notal Vision Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: C2021.002
Record Dates: First submitted 2022-03-06; First posted 2022-03-15 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-02

CONDITIONS: Neovascular Age-related Macular Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study will enroll up to 30 AMD patients diagnosed with NV-AMD in at least one eye at the time of enrollment. At the Study Visit, fluid must be present in at least one eye of the subjects. If only one eye qualifies for enrollment, that will be assigned as the study eye. If both eyes are eligible, the study eye will be assigned according to a randomization schedule. Only one eye of each subject will be enrolled in the study. All subjects will be enrolled at 1 site in the United States. Subjects must meet all inclusion and no exclusion criteria.

DETAILED DESCRIPTION:
Description of Study Procedures and In-Office Visit:

Enrollment/Screening:

At the Enrollment/ Screening Visit, the exams will be conducted in the following order:

1. Patient will be informed concerning the study and sign the Informed Consent Form (ICF) prior to conduct of any study procedures.
2. The following data will be collected for each study subject:

   1. Subject's DOB
   2. Gender
   3. Number and type of injections and last injection date
3. The following data will be collected for the study eye:

   1. Qualifying diagnosis for the study eye from the subject's medical record
   2. From the subject's medical record, the presence of other ophthalmic conditions including but not limited to:

   i. Cataract ii. Glaucoma iii. Dry Eye iv. Other macula findings, e.g., epi retinal membrane, macular hole, vitreo-macular traction (VMT)
4. Refraction correction
5. Snellen BCVA on both eyes on the day of the visit.
6. Selecting the study eye:

   1. Both eyes of the subject will be scanned, non-dilated, with a Zeiss Cirrus OCT device to get an acceptable single volume scan per eye. Scanning pattern to be used: Macular cube, 6X6mm, 128 B-scans per volume scan
   2. The PI/CoPI will read the Zeiss Cirrus OCT scans of both eyes and will grade each eye for the presence/absence of SRF and/or IRF in the retina
   3. The eye with SRF and/or IRF will be set as the study eye. In case both eyes were graded as fluid-present, the study eye will be set randomly
   4. The Zeiss Cirrus OCT scan of the study eye will be part of the study analysis

NOTE: Any planned treatment for NV-AMD should be administered after completion of all study-related scans

OCT Scans:

1. The study eye of the subject will be scanned once, non-dilated, with a Zeiss Cirrus OCT device to get an acceptable single volume scan of the study eye in each repetition.

   Scanning pattern to be used: Macular cube, 6X6mm, 128 B-scans per volume scan
2. Following the Zeiss Cirrus OCT scans, the subject will be placed in a room with the Notal OCT V3.0 device which has been set up by a technician.
3. Notal OCT V3.0 scans

   1. The technician will register the subject using the touchscreen of the Notal OCT V3.0 device and the assigned Subject ID.
   2. On the first Notal OCT V3.0 device the subject will perform a self-tutorial.
   3. The technician will set the first Notal OCT V3.0 for self-scan of the study eye. The subject will perform the tutorial on the eye with better vision, based on the subject's subjective decision, even if that eye is not the study eye. Then, the subject will perform on the first device- a calibration, and 5 volume scans.
   4. The technician will set the second device for self-scans of the study eye. The subject will perform calibration and 5 volume scans.
   5. The subject will be able to rest 1-2 minutes between self-scans
4. Collect AEs, if applicable.
5. Exit the subjects from the study.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to speak, read and understand English.
2. Ability to understand and agree to contents of informed consent in writing or verbal.
3. Adult diagnosed with NV-AMD in at least one eye based on the subject's medical record.
4. Fluid presence in the study eye per the PI review of Screening commercial OCT.
5. Best corrected Visual Acuity of 20/320 or better in the study eye.
6. Available and willing to conduct self-scanning in the office

Exclusion Criteria:

1. Any other retinal disease requiring steroidal or anti-VEGF injections.
2. Dilated pupils

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 30 AMD patients diagnosed with NV-AMD in at least one eye at the time of enrollment. At the Study Visit, fluid must be present in at least one eye of the subjects. If only one eye qualifies for enrollment, that will be assigned as the study eye. If both eyes are eligible, the study eye will be assigned according to a randomization schedule. Only one eye of each subject will be enrolled in the study. All subjects will be enrolled at one 1 site in the United States.
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2021-09-13 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2022-01-05 (Actual)

PRIMARY OUTCOMES:
Notal Home OCT Total Retinal Fluid (TRF) amount measured by NOA | 5 minutes
  volume [nl] of the TRF
Notal Home OCT Intra-Retinal Fluid (IRF) amount measured by NOA | 5 minutes
  volume [nl] of the IRF
Notal Home OCT Sub-Retinal Fluid (SRF) amount measured by NOA | 5 minutes
  volume [nl] of the SRF
Zeiss Cirrus OCT Total Retinal Fluid (TRF) amount measured by a human reader | 5 minutes
  volume [nl] of the TRF
Zeiss Cirrus OCT Intra-Retinal Fluid (IRF) amount measured by a human reader | 5 minutes
  volume [nl] of the IRF
Zeiss Cirrus OCT Sub-Retinal Fluid (SRF) amount measured by a human reader | 5 minutes
  volume [nl] of the SRF

SECONDARY OUTCOMES:
Subjects who completed self-scanning on the Notal Home OCT, following a self-tutorial. | 5 minuts
  Number of subjects and percentage of subjects who completed self-scanning on the Notal Home OCT, following a self-tutorial.

CONTACTS AND LOCATIONS:
Overall Officials: Gidi Benyamini, Study Chair — Notal vision Druyanov 5, Tel Aviv
Locations (1):
- Elman Retina Group, Glen Burnie, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided